CLINICAL TRIAL: NCT03256201
Title: Preoperative Exercise and Nutrition to Improve Pancreatic Cancer Outcomes by Targeting Sarcopenia: A Translational Pilot RCT
Brief Title: Exercise and Nutrition to Improve Pancreatic Cancer Outcomes
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Oklahoma (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: 5991
Record Dates: First submitted 2017-05-26; First posted 2017-08-21 (Actual); Last update posted 2024-08-16 (Actual); Status verified 2024-08

CONDITIONS: Pancreatic Cancer
Keywords: Cancer; prehabilitation; sarcopenia
MeSH Terms: conditions — Pancreatic Neoplasms; Neoplasms; Sarcopenia | interventions — Nutrition Assessment

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Standard Exercise Group (Experimental): Patients receive a single instruction session with a physical therapist, for training in moderate intensity (using Rate of Perceived Exertion) exercise including cardiovascular endurance, flexibility, and AROM of upper and lower body. If no other preferred mode of endurance training, a home ergometer is provided for use with arms and/or legs.
  Interventions: Behavioral: Nutritional Counseling; Behavioral: Standard Exercise
- Enhanced Exercise Group (Experimental): Patients receive a single instruction session with a physical therapist, for training in moderate intensity (using Rate of Perceived Exertion) exercise including cardiovascular endurance, flexibility, and resistance exercise for upper and lower body. If no other preferred mode of endurance training, a home ergometer is provided for use with arms and/or legs.
  Interventions: Behavioral: Nutritional Counseling; Behavioral: Enhanced Exercise

INTERVENTIONS:
Behavioral: Nutritional Counseling — Patients in both arms receive a single counseling session with a licensed dietician to determine individual protein goal for body weight and current dietary intake. Goal is then met through protein supplementation (provided) if needed beyond dietary intake.
Behavioral: Standard Exercise — Patients receive a single instruction session with a physical therapist, for training in moderate intensity (using Rate of Perceived Exertion) exercise including cardiovascular endurance, flexibility, and AROM of upper and lower body. If no other preferred mode of endurance training, a home ergometer is provided for use with arms and/or legs.
  Arms: Standard Exercise Group
Behavioral: Enhanced Exercise — Patients receive a single instruction session with a physical therapist, for training in moderate intensity (using Rate of Perceived Exertion) exercise including cardiovascular endurance, flexibility, and resistance exercise for upper and lower body. If no other preferred mode of endurance training, a home ergometer is provided for use with arms and/or legs.
  Arms: Enhanced Exercise Group

SUMMARY:
This is a blinded pilot study in which patients scheduled for pancreaticoduodenectomy for pancreatic or related cancers are randomized to dietary counseling and home exercise at high weekly frequency, either with or without individualized resistance training, in order to determine if such an intervention and research design are feasible in this population. We also aim to determine if physical function or quality of life can be improved with only 2-3 weeks of prehabilitation. This is in preparation for a larger study to determine if resistance improves outcomes.

DETAILED DESCRIPTION:
This initial feasibility and proof of concept study focuses on maximizing pancreatic cancer survivors' fitness and physical function in a brief period, the 2-3 weeks available prior to surgical resection, using a home-based exercise program with all equipment provided, and following nutritional recommendations. Intervention begins when the oncologist determines that the patient is a candidate for pancreaticoduodenectomy, and continues until surgery. Participants in both arms are asked to perform moderate exercise daily, targeting a total of 60 minutes per day by the surgery date, but in bouts as short as a few minutes each, and progressed according to tolerance. Initial prescription is individualized according to the patient's baseline level of exercise and functional status. Patients record their exercise and wear an accelerometer to track activity if willing. All participants receive follow-up phone calls from an exercise specialist for adherence and assistance with progression. The intervention period ends at the time of surgery.

In this 'quasi-double blinded' randomized trial, participants are not told the difference between the two exercise interventions, and randomization to the two treatment arms is stratified by baseline functional status, such that patients deemed to be 'borderline' in fitness for surgery are distributed across the groups. Prior chemotherapy exposure is allowed and recorded.

ELIGIBILITY:
Inclusion:

* Individuals with suspected pancreatic or related tumor for surgical resection by pancreaticoduodenectomy, including those who've received neoadjuvant chemotherapy, are eligible provided they are approved for exercise participation by pancreatic clinic team.
* Cognition and English language skills must be sufficient for completion of consent and questionnaires.
* Age >30.
* Able to rise from a chair and walk household distances without assist from another person.
* Willing to be randomized to one of two pre-operative home-based exercise programs, without knowing the difference between the two, and use protein supplementation if instructed.

Exclusion:

* Individuals are excluded if they are unsafe (according to the study team) based on current MD recommendation not to exercise, medical history, recent fracture or high-risk bone lesion, or neurologic disorder with safety concerns.
* Participants cannot have an allergy to whey protein, or abnormal response to baseline physical performance tests of walking endurance and strength.
* Those who currently participate in a regular and substantial (as defined by the study team) strengthening or protein supplementation program are eligible only for the 'for assessment only' observational version of the study, but will not be included in the randomized trial.

Min Age: 30 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 95 (Actual)
Dates: Start 2016-02-01 (Actual); Primary Completion 2024-04-01 (Actual); Study Completion 2025-03 (Estimated)

PRIMARY OUTCOMES:
Accrual | 2 year
  The percentage of eligible patients enrolled
Retention | 2 year
  Retention as the percentage of enrolled patients retained assessment point
Adherence | 2 year
  Adherence will be estimated as percentage of prescribed exercise completed based on exercise diaries and phone calls

SECONDARY OUTCOMES:
Quality of Life Assessment | Approximately 1-3 days pre-op
  Quality of life will be assessed using Functional Assessment of Cancer Therapy General Scale (FACT-G) during the pre-operative period (V1-V2). Scale is 0-108. The higher the score, the better the score.
Change in Body Weight | Approximately 1-3 days pre-op
  Change in baseline body weight in pounds during the pre-operative period (V1-V2)
Change in Body Weight | Approximately 1-3 days pre-op
  Change in baseline body weight in pounds at second post operative visit
Physical Performance | Approximately 1-3 days pre-op
  Six-Minute Walk Test in meters during the pre-operative period (V1-V2). The Six Minute Walk test will be performed according to American Thoracic Society Guidelines.
Physical Performance | Approximately 2-4 weeks pre-op
  Gait Speed at usual pace
Physical Performance | Approximately 1-3 days pre-op
  Grip Strength . with a Jamar handgrip dynamometer .
Physical Performance | Approximately 4 months post-op
  Sit-to-Stand .Time to 5th Stand will be performed according to the Short Performance Physical Battery.
Assessment of Symptoms | Approximately 4 weeks post-op
  Functional Assessment of Cancer Therapy - Hepatobiliary (FACT-Hep), at first post-operative visit.
Assessment of Symptoms | Approximately 1-3 days pre-op
  Functional Assessment of Anorexia-Cachexia Therapy - FAACT, during the pre-operative period (V1-V2).

CONTACTS AND LOCATIONS:
Overall Officials: Elizabeth Hile, PhD, PT, Principal Investigator — Faculty
Locations (1):
- University of Oklahoma Health Sciences Center, Oklahoma City, Oklahoma, United States

IPD SHARING:
Plan to Share IPD: No